CLINICAL TRIAL: NCT07336966
Title: Does Recessive Optic Atrophy Due to WFS1 is a Specific Entity Different From Wolfram Syndrome?
Brief Title: Does Recessive Optic Atrophy Due to WFS1 Exist?
Status: Not yet recruiting | Type: Observational
Sponsor: Hôpital Necker-Enfants Malades (Other)
Responsible Party: Principal Investigator, Christophe Orssaud, MD, Responsible CRMR Ophtara HEGP, European Georges Pompidou Hospital
Other Study IDs: ROAWFS1
Record Dates: First submitted 2025-11-15; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Wolfram Syndrome 1; Optic Atrophies, Hereditary
Keywords: WFS1; Wolfram syndrome; hereditary optic neuropathy
MeSH Terms: conditions — Wolfram Syndrome; Optic Atrophies, Hereditary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- wolfram syndrome: Patients according to the EuroWABB criterions of Wolfram syndrome and French national guidelines
  Interventions: Other: analyse study
- recessive optic atrophy: patients with an OA due to mutation of gene WFS1, whatever its age of occurrence, without any other clinical manifestation.
  Interventions: Other: analyse study

INTERVENTIONS:
Other: analyse study — Retrospective analyse and study of recorded data of patients with wolfram syndrome or recessive optic atrophy due to WFS1 mutation

SUMMARY:
All patients with Wolfram syndrome and recessive optic atrophy due to a mutation of the WFS1 from a single Center were included in a retrospective study. Evolution of the visual acuity since the occurrence of the optic atrophy and its last value, OCT data, genetic data and systemic manifestations were analyzed.

DETAILED DESCRIPTION:
Ophthalmological date will be include : farsighted best corrected visual acuity (BCVA) assessment, slit-lamp examination of the anterior segment, Goldman aplanation tonometry, funduscopy, retinography, Goldman manual visual field and optical coherent tomography (OCT). These will include global value of Retinal Nerve Fiber Layer (RNFL) thickness as well as the ganglion cell complex (GCC) thickness.

ELIGIBILITY:
Inclusion Criteria:

* WFS1 mutation

Exclusion Criteria:

* WFS2 mutation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient from our rare disease reference center
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Visual acuity at the last visit | The last visit will be registered regardless of the time elapsed since the onset of the disease, considered as a baseline
  Comparison of visual acuity at the last visual between the 2 groups

SECONDARY OUTCOMES:
Evolution of visual acuity | Measurement at the occurence of the disease considered as baseline and at the last visit
  We only take in account the first visual assessments and the delay from the occurrence of the OA as well as the last visual assessment when possible and the delay between those two examinations.
Age | At the occurence of the disease considered as baseline
  Age of the patient at the occurrence of the disease
Global RNFL thickness | Measurement at the occurence of the disease considered as baseline and at the last visit
  Comparison of the global RNFL thickness according to the group and delay from occurence of the disease

IPD SHARING:
Plan to Share IPD: No